CLINICAL TRIAL: NCT03781544
Title: Effect of Opioids and NSAIDs on Sympathetic Nervous System and Vascular Function in Healthy Subjects and Patients With Osteoarthritis
Brief Title: Effects of Opioids and NSAIDs on Sympathetic Nervous System and Vascular Function
Acronym: OPIOVASC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPIOVASC
Record Dates: First submitted 2018-12-03; First posted 2018-12-20 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis of Multiple Joints of Ankle or Foot; Healthy
MeSH Terms: interventions — Tramadol; Acetaminophen; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diclofenac (Experimental): Diclofenac (Diclofenacum natricum) A single i.v. infusion of Diclofenac (dose: 75mg/100ml) will be administered to the participants (treatment arm).
  Interventions: Drug: Diclofenac
- Paracetamol (Active Comparator): Paracetamol (Paracetamol Sintetica):
  A single i.v. infusion of Paracetamol (dose: 1g/100ml) will be administered to the participants (control arm).
  Interventions: Drug: Paracetamol
- Tramadol (Experimental): Tramadol (Tramadol-Mepha):
  A single i.v. infusion of Tramadol (dose: 400mg/100ml) will be administered to the participants (treatment arm).
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Tramadol — A single i.v. infusion of Tramadol (dose: 400mg/100ml) will be administered to the participants (treatment arm).
  Other Names: Tramadol-Mepha
  Arms: Tramadol
Drug: Paracetamol — A single i.v. infusion of Paracetamol (dose: 1g/100ml) will be administered to the participants (control arm).
  Other Names: PARACETAMOL Sintetica
  Arms: Paracetamol
Drug: Diclofenac — A single i.v. infusion of Diclofenac (dose: 75mg/100ml) will be administered to the participants (treatment arm).
  Arms: Diclofenac

SUMMARY:
Evaluation of the effect of different analgesic treatments (Tramadol, Paracetamol, Diclofenac) on sympathetic nerve activity, blood pressure, heart rate, heart rate, and vascular function in osteoarthritis patients and healthy subjects.

DETAILED DESCRIPTION:
Hundreds of millions of patients worldwide require pain-relieving therapy to maintain an acceptable quality of life. Pain relievers, including non-steroidal anti-inflammatory drugs (NSAIDs) and opioids, however, exert unwanted potent adverse systemic off-target effects and their use is associated with a well-documented excess of cerebrovascular and cardiovascular events. This of particular concern for the one fourth of the world's population aged over 35 years suffering from chronic pain, particularly with arthritis of whom half also present with established or at high risk of cardiovascular disease. This uncertainty around the cardiovascular safety of pain relieving drugs leaves practitioners and their patients with difficult management decisions and underscores the need to investigate potential differential cardiovascular effects of NSAIDs and opioids and to better delineate the underlying mechanisms involved. Indeed, currently available NSAIDs invariably disrupt the balance between prostacyclin and thromboxane, but may also exert multiple and opposing cardiovascular effects on endothelial factors, including nitric oxide and reactive oxygen species, the sympathetic nervous system and vascular inflammation. Intriguingly, the net effect of pain relieving drugs on vascular function and sympathetic nerve activity and its resulting deterioration of blood pressure control is increasingly recognized as a major possible determinant in explaining the cardiovascular side effects of NSAIDs. As a result of the ongoing concerns around the cardiovascular safety of NSAIDs and coxibs many patients are being withheld effective pain relieve or switched to opioids and/or paracetamol under the assumption of their yet unproven greater cardiovascular safety. The absence of evidence about the cardiovascular safety of these drugs presents a major dilemma for patients and physicians, who have been warned about the toxicity of NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age, male or female, with a diagnosis of osteoarthritis or healthy subjects ≥ 18 years of age;
2. Written informed consent;

Exclusion criteria:

1. History of hypersensitivity or allergy to any of the study drugs
2. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or other major CV surgery, percutaneous coronary intervention (PCI) or carotid angioplasty within the 3 months prior to Visit 1;
3. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within the 3 months after Visit 1;
4. Presence of significant endocrine diseases;
5. Presence of active acute infectious diseases;
6. Known narrow-angle glaucoma;
7. Known epilepsy;
8. Cimino-shunt operation on both arms;
9. Pregnancy, intention thereof during study, lack of sufficient contraception, breastfeeding;
10. Drug or alcohol abuse;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
resting MSNA (sympathetic nervous activity ) | 1day (110 min)
  Effect of different single analgesic treatments (Tramadol, Paracetamol, Diclofenac) on resting muscle sympathetic nerve activity (MSNA) in osteoarthritis patients (post 2 days of analgesic therapy washout phase) and in healthy subjects.
  Tramadol treatment will be compared to diclofenac and paracetamol (3 treatment arms).
  90 participants (45 osteoarthritis patients, 45 healthy subjects);
  Single infusion of Tramadol (50 mg i.v.) Single infusion of Paracetamol (1000 mg i.v.) Single infusion of Diclofenac (75 mg i.v.)
changes in FMD (Flow mediated vasodilation) | 1 day (210min)
  Effect of a single acute intravenous analgesic treatment with tramadol versus paracetamol on changes in flow mediated dilatation (FMD) in osteoarthritis patients and in healthy subjects.
  Tramadol treatment will be compared with paracetamol as we previously demonstrated that paracetamol exerts no significant effects on endothelial function as measured by flow mediated dilatation.
  80 participants (40 osteoarthritis patients, 40 healthy subjects);
  Single infusion of Tramadol (50 mg i.v.) Single infusion of Paracetamol (1000 mg i.v.)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ruschitzka, MD, Study Director — Cardiology, University Heart Center Zurich
Locations (1):
- University Heart Center Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No